CLINICAL TRIAL: NCT01964027
Title: The Study of Irinotecan Plus Epirubicin as the Second-line Chemoregime for Advanced Gastric Cancer
Acronym: SIEG
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Pan Yueyin, Professor, Anhui Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIEG
Record Dates: First submitted 2012-01-19; First posted 2013-10-17 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2013-10

CONDITIONS: Stage IV Gastric Cancer With Metastasis
Keywords: second line chemoregime; gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Irinotecan; Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Irinotecan plus epirubicin (Experimental): Irinotecan(Camptosar)150mg /m2 d1,（intravenous infusion of 30-90 minutes) + epirubicin(Pharmorubicin) 50mg/m2 (total dose does not exceed 700mg/m2) every 21days for 1 treatment * 6 cycles as the second line chemoregime for advanced gastric cancer
  Interventions: Drug: second line chemoregime for advanced gastric cancer

INTERVENTIONS:
Drug: second line chemoregime for advanced gastric cancer — Irinotecan(Camptosar)150mg /m2 d1,（intravenous infusion of 30-90 minutes) + epirubicin(Pharmorubicin) 50mg/m2 (total dose does not exceed 700mg/m2) every 21days for 1 treatment * 6 cycles as the second line chemoregime for advanced gastric cancer
  Other Names: irinotecan plus epirubicin

SUMMARY:
This study is to determine the response rate and safety profile of irinotecan plus epirubicin as the second-line chemotherapy for advanced gastric cancer and fully evaluate the feasibility and effectiveness of the regime.

DETAILED DESCRIPTION:
The main purposes: to determine the progression-free survival (PFS) and overall survival (OS) of gastric cancer patients given irinotecan + epirubicin as second-line treatment, who are at Stage IV with disease progressed or recurred after first-line chemotherapy failed, ,

The Secondary purposes: to determine disease control rate (Disease Control Rate, DCR), the objective response rate (Object Response rate, ORR) and the Quality of life (Quality Of Life, QOL)

ELIGIBILITY:
Inclusion criteria:

* Aged between 18 to 70 years
* The pathologically confirmed gastric adenocarcinoma and the failure of first-line chemotherapy
* Measurable lesions outside the stomach
* ECOG(Eastern Cooperative Oncology Group ) score between 0 to 1
* Expected survival time of at least 3 months
* Subjects receiving treatment for other damage caused has been restored, which it accepted the nitroso or mitomycin interval> 6 weeks, the acceptance of other cytotoxic drugs, radiotherapy or surgery> = 4 weeks, and the wound has completely healed. No bleeding, no nervous system transferred
* Blood and organ function was normal

Exclusion criteria:

* Comorbid with other malignant tumors
* Pregnant and lactating women
* with the disease of endangering patient's safety and affecting the completion of the study
* Patients suffering from high blood pressure by antihypertensive treatment cannot control (systolic blood pressure> 140mmhg, diastolic blood pressure> 90mmhg,) there is more than Class I and Class I arrhythmia coronary heart disease, with more than Class I heart dysfunction
* Major organ failure, such as decompensated heart and lung failure, liver failure, renal failure and patients with intestinal obstruction ipate in other clinical trials of patients in the past four weeks
* Participated in clinical trials with other drugs or using other drugs during past 4 weeks
* Lesions which can't be measured such as pleural effusion, ascites, peritoneal cancer lesions, diffuse liver and bone metastases violation, brain metastasis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-07 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
PFS and OS | 2 years
  Evaluation progression-free survival (PFS) and overall survival (OS)
  RECIST(Response Evaluation Criteria In Solid Tumors)1.1:
  1. Complete response (CR)
  2. Partial response (PR)
  3. Stable disease(SD) and progression disease(PD)
  4. CR + PR is efficient.

CONTACTS AND LOCATIONS:
Overall Officials: Yueyin Pan, MD, Principal Investigator — The First Affiliated Hospital of Anhui Medical University
Locations (1):
- Department of Oncology,The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China